CLINICAL TRIAL: NCT00117494
Title: Randomised Comparative Study of the Efficacy and Safety of Rosuvastatin and Pravastatin in Dyslipidemic Patients Treated With Antiretroviral Agents. Anrs 126
Brief Title: Rosuvastatin Versus Pravastatin in HIV Patients Treated With Boosted Protease Inhibitors (PI) (ANRS126)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001451-38; ANRS 126
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Hyperlipidemia; HIV Infections
Keywords: Hyperlipidemia; HIV infections; STATINS, HMG-COA; Protease Inhibitor; Treatment Experienced
MeSH Terms: conditions — Hyperlipidemias; HIV Infections | interventions — Pravastatin; Rosuvastatin Calcium

INTERVENTIONS:
Drug: Pravastatin
Drug: Rosuvastatin

SUMMARY:
In HIV hypercholesterolemic patients treated with protease inhibitors, some drugs of the statin group are used to control cholesterol level. New and potentially more efficient statins may interfere with protease inhibitors and hence loose a part of their activity. They have thus to be compared with a more established drug of the same class (e.g. pravastatin). The protocol compares the efficacy and safety of rosuvastatin and pravastatin.

DETAILED DESCRIPTION:
The study compares the efficacy and safety of rosuvastatin and pravastatin among dyslipidemic HIV-seropositive patients treated with antiretroviral agents including a boosted protease inhibitor.

It is an open, multicenter, randomised trial, with two parallel groups comparing rosuvastatin with pravastatin.

Statins are administered from D0, with a single daily dose in the morning, for 45 consecutive days.

The duration of the study for each patient will be 45 days not including the preselection period (maximum 15 days).

The primary end-point compares the change in LDL cholesterol between D0 and D45, in patients receiving rosuvastatin (10 mg/day) or pravastatin (40 mg/day) and treated by antiretroviral agents including a boosted Protease Inhibitor.

Secondary end-points compares changes in triglycerides and HDL cholesterol; percentage of patients with a normal value of LDL cholesterol, HDL cholesterol and triglycerides on D45; clinical safety and laboratory safety parameters of rosuvastatin and pravastatin; distribution profile of the diameter of LDL cholesterol particles.

Cmin of rosuvastatin, pravastatin and protease inhibitors (PI) are controlled at D15 for statins and PI.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL cholesterol over 4.1 mmol/L (1.6 g/l)
* Blood triglycerides over 8.8 mmol/L (8 g/l)
* HIV-1 infection
* Viral load above or equal to 10.000 copies/ml
* Stable antiretroviral regimen for past two months

Exclusion Criteria:

* Coronary disease
* Genetic muscular disease
* CPK over 5N
* Hepatic or renal insufficiency
* Alcohol intake more than 40g/d
* Hypothyroidism
* Pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Compare the change in LDL cholesterol between D0 and D45, in patients receiving rosuvastatin (10 mg/day) or pravastatin (40 mg/day) and treated by antiretroviral agents including a boosted protease inhibitor on D45.

SECONDARY OUTCOMES:
Changes in triglycerides and HDL cholesterol on D45
Percentage of patients with a normal value of LDL cholesterol, HDL cholesterol and triglycerides on D45 Clinical and biological safety parameters of rosuvastatin and pravastatin
Distribution profile of the diameter of LDL cholesterol particles
Cmin of rosuvastatin and pravastatin on D15
Cmin of protease inhibitors on D15.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Aslangul, MD, Principal Investigator — Hopital Hôtel Dieu Paris; Dominique Costagliola, Study Director — Inserm U720 Paris Pitié Salpétrière
Locations (1):
- service de Médecine Interne Hopital Hotel Dieu, Paris, France

REFERENCES:
- [Derived] Bittar R, Giral P, Aslangul E, Assoumou L, Valantin MA, Kalmykova O, Federspiel MC, Cherfils C, Costagliola D, Bonnefont-Rousselot D; French National Agency for AIDS and Viral Hepatitis Research (ANRS) 126 study group. Effects of rosuvastatin versus pravastatin on low-density lipoprotein diameter in HIV-1-infected patients receiving ritonavir-boosted protease inhibitor. AIDS. 2012 Sep 10;26(14):1801-5. doi: 10.1097/QAD.0b013e328357063c. PMID 22739396
- [Derived] Bittar R, Giral P, Aslangul E, Assoumou L, Valantin MA, Kalmykova O, Fesel-Fouquier V, Costagliola D, Bonnefont-Rousselot D; ANRS 126 study group. Determinants of low-density lipoprotein particle diameter during antiretroviral therapy including protease inhibitors in HIV-1-infected patients. Antivir Ther. 2012;17(5):855-60. doi: 10.3851/IMP2065. Epub 2012 Feb 9. PMID 22318219